CLINICAL TRIAL: NCT03651349
Title: A Phase I Study to Determine the Maximum Tolerated Dose (MTD) of HK-001 and to Evaluate Its Pharmacokinetic Profile in Healthy Volunteers
Brief Title: To Determine the Maximum Tolerated Dose (MTD) of HK-001 in Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Everfront Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFBORAZ20141120
Record Dates: First submitted 2018-08-26; First posted 2018-08-29 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Placebo control (Placebo Comparator): Eligible subjects will receive either different dosages of HK-001 or placebo in a 3:1 ratio in 1 of the 7 dose cohorts consisting of 8 subjects each.
  Interventions: Drug: Placebo control
- 50 mg, BID (Experimental): Eligible subjects will receive either different dosages of HK-001 or placebo in a 3:1 ratio in 1 of the 7 dose cohorts consisting of 8 subjects each.
  Interventions: Drug: HK-001
- 100 mg, BID (Experimental): Eligible subjects will receive either different dosages of HK-001 or placebo in a 3:1 ratio in 1 of the 7 dose cohorts consisting of 8 subjects each.
  Interventions: Drug: HK-001
- 150 mg, BID (Experimental): Eligible subjects will receive either different dosages of HK-001 or placebo in a 3:1 ratio in 1 of the 7 dose cohorts consisting of 8 subjects each.
  Interventions: Drug: HK-001
- 225 mg, BID (Experimental): Eligible subjects will receive either different dosages of HK-001 or placebo in a 3:1 ratio in 1 of the 7 dose cohorts consisting of 8 subjects each.
  Interventions: Drug: HK-001
- 300 mg, BID (Experimental): Eligible subjects will receive either different dosages of HK-001 or placebo in a 3:1 ratio in 1 of the 7 dose cohorts consisting of 8 subjects each.
  Interventions: Drug: HK-001
- 400 mg, BID (Experimental): Eligible subjects will receive either different dosages of HK-001 or placebo in a 3:1 ratio in 1 of the 7 dose cohorts consisting of 8 subjects each.
  Interventions: Drug: HK-001
- 525 mg, BID (Experimental): Eligible subjects will receive either different dosages of HK-001 or placebo in a 3:1 ratio in 1 of the 7 dose cohorts consisting of 8 subjects each.
  Interventions: Drug: HK-001

INTERVENTIONS:
Drug: HK-001 — HK-001 is synthesized by PharmaCore Biotech Co., Ltd. Synthetic (Z)-BP with high purity will be used in this proposed study.
  Other Names: (Z)-n-butylidenephthalide [(Z)-BP]
  Arms: 100 mg, BID; 150 mg, BID; 225 mg, BID; 300 mg, BID; 400 mg, BID; 50 mg, BID; 525 mg, BID
Drug: Placebo control — In order to evaluate the safety and tolerability of HK-001 more accurately, a drug-free placebo control is planned to be utilized for the same administration route in this proposed trial. The placebo control that is identical in appearance, smell, weight, and excipients will be supplied by Everfront Biotech Inc.
  Other Names: Placebo
  Arms: Placebo control

SUMMARY:
Eligible subjects will receive either different dosages of HK-001 or placebo in a 3:1 ratio in 1 of the 7 dose cohorts. After single dose administration, followed by an independent Data and Safety Monitoring Board (DSMB) meeting for safety assessments (including the available plasma pharmacokinetic profile), the subjects will be allowed to receive (Z)-BP or placebo twice a day orally at the study site for 14 consecutive days and follow up on the 28th day after the last dose administration by a site visit. The study drugs (including placebo) will be administered at the study site by following the investigator's instructions to either perform blood sampling for pharmacokinetic evaluation or maximize the treatment compliance.

There will be 7 cohorts and subjects will be randomized into cohorts consisting of 8 subjects each (6 active and 2 placebo controls per cohort). Dose cohorts will be escalated sequentially from low to high dose (50 mg, BID; 100 mg, BID; 150 mg, BID; 225 mg, BID; 300 mg, BID; 400 mg, BID; 525 mg, BID) by following a modified Fibonacci sequence, and based on the decision of an independent DSMB at a set time point. Following all subjects of a cohort complete the safety and PK evaluation after receiving the last dose administration, a cohort at the next dose level will be launched if the DSMB does not identify significant safety concerns after reviewing safety data and PK profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age is no less than 20 years old.
2. Subjects whose body mass index (BMI) at screening is within a range of ≥18.5 kg/m2 and <25.0 kg/m2.

   BMI = Body Weight (kg) / [Height (m)]2 And body weight is not less than 50 kg and 45 kg for males and females, respectively.
3. Subject's medical history shows no contraindication to the test medications [hypersensitivity to (Z)-BP or any component of test and reference products].
4. Subjects who are judged to be in good health by the investigator based upon the results of physical examinations (PEs) and chest X-ray (within 60 days prior to the first study dose), and all items of routine laboratory tests, including serum biochemistry, hematology and urinalysis, are within normal range as judged by the site. Assessment items of blood biochemistry include electrolytes (sodium, potassium, chloride, calcium, phosphorus), albumin, total cholesterol, total bilirubin, ALP, SGOT, SGPT, GGT, BUN, PT, APPT, serum creatinine, triglyceride, glucose, amylase, lipase, ACTH, aldosterone, cortisol, T3, free T4, TSH, and uric acid. Assessment items of hematology tests include red blood cell (RBC), white blood cell (WBC) and platelet count; differential WBC count including neutrophils, lymphocytes, monocytes, eosinophils, and basophils; hemoglobin, and hematocrit. Assessment items of urinalysis include appearance, gravity, pH, erythrocyte, leukocyte, epithelial cells, glucose, protein, ketones, and nitrite
5. Female subjects show negative pregnancy test results within 30 days prior to the first study dose.
6. Subjects did not take any of the following medications in the specified durations:

   * Any medication (except contraceptives) within 14 days prior to the first dose of the study
   * Any enzyme inducer or inhibitor within 30 days prior to the first dose of the study
7. Subjects understood and have signed the written informed consent form.

Exclusion Criteria:

1. Subjects with any properly diagnosed disease within 30 days prior to the first dose of the study
2. Subjects with a clinically significant hematological, endocrinal, cardiovascular, hepatic, renal, gastrointestinal, and/or pulmonary disorders; subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism and excretion of drugs; subjects who have had any previous gastrointestinal surgery, except appendectomy if performed >90 days prior to the first dose of the study
3. Subjects who have received any known hepatic or renal clearance-altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazine, clarithromycin, trolearndomycin, ketoconazole, miconazolem fluconazole, itraconazole) for a period of up to 30 days prior to the first dose of the study
4. Subjects had participated in investigational drug trials and took any investigational drugs within 60 days prior to the first study dose.
5. Subjects had blood donation for more than 250 mL within 60 days prior to the first dose of the study.
6. Subjects had a history of drug abuse or alcohol abuse according to DSM IV criteria.
7. Subjects who are smokers or have smoking history
8. Subjects who cannot stop caffeine-intakes for 48 hours prior to the first study dose and during the entire study period.
9. Subjects who are pregnant or lactating
10. For enrollment of female subjects with child-bearing potential, the subject must be practicing sexual abstinence or be using and willing to continue to use a medically acceptable form of birth control for at least 1 month prior to screening (that period will extend to 3 months for oral contraceptive use) and for at least 30 days after the last dose of study drug. For a subject to be considered not to be of child-bearing potential, she must have been amenorrheic for at least 2 years, or must have had a hysterectomy, a bilateral tubal ligation, and/or a bilateral oophorectomy (as determined by the medical history). The male partner of a female study subject with childbearing potential must use a condom and ensure that his partner uses a suitable method of contraception as outlined above.
11. Subjects who are inappropriate to participate in this study, as judged by the clinical investigator
12. Subjects who have been tested positive for the following tests:

    * Human immunodeficiency virus (HIV)
    * Hepatitis B virus (HBV)
    * Hepatitis C virus (HCV)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 48 days
  The MTD will be determined by study definition as the highest dose level without significant safety and tolerability concern.
Dose Limiting Toxicities (DLT) | 48 days
  In this study, the DLTs are defined as below:
  1. Any Grade ≥2 AE found during study period that is considered at least possibly drug related as judged by the investigator. The NCI-CTCAE 4.03 will be used to grade serum chemistry, hematology, and other abnormalities in the current study.
  2. Any drug-related (including probably or possibly drug-related) serious adverse event (SAE) found during study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No